CLINICAL TRIAL: NCT06362109
Title: The Impact of Intermittent Nutritional Tube Supplementation in Elderly Patients With Dysphagia: A Randomized Controlled Study
Brief Title: The Impact of Intermittent Nutritional Tube Supplementation in Elderly Patients With Dysphagia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhao Song Ling (Other Government)
Responsible Party: Sponsor-Investigator, Zhao Song Ling, Research Director, Chest Hospital, Ministry of Health and Welfare, Taiwan
Organization: Chest Hospital, Ministry of Health and Welfare, Taiwan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Once tubefeeding
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine rehabilitation group (Active Comparator): This group is going to receive Routine rehabilitation once a day.
  Interventions: Behavioral: Routine rehabilitation
- Routine rehabilitation + Intermittent Oro-esophageal Tube Feeding group (Experimental): This group is going to receive Routine rehabilitation once a day and Intermittent Oro-esophageal Tube Feeding once a day.
  Interventions: Behavioral: Routine rehabilitation; Device: Intermittent Oro-esophageal Tube Feeding

INTERVENTIONS:
Behavioral: Routine rehabilitation — Routine rehabilitation consists of:
  1. Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  2. Swallowing training, including lemon ice stimulation, empty swallowing training, and pronunciation training.
  3. Pulmonary function training, including standing training, cough training, and diaphragm muscle training.
Device: Intermittent Oro-esophageal Tube Feeding — The group is given enteral nutritional support with Intermittent Oro-esophageal Tube according to the following procedure: Before each feeding, inside and outside of the tube was cleaned with water. During feeding, the patient should maintain a semi-reclining or sitting position with mouth opened, and the tube was inserted slowly and smoothly into the upper part of the esophagus by medical staffs while the appropriate depth of intubation was checked with the calibration markings on the tube wall. The distance from the incisors to the head part of the tube should be between 22-25 cm.
  Arms: Routine rehabilitation + Intermittent Oro-esophageal Tube Feeding group

SUMMARY:
This is a prospective, randomized controlled clinical trail involved Elderly Patients With Dysphagia.The goal of this clinical trial is to compare the clinical effect of Intermittent Oro-esophageal Tube Feeding in Elderly Patients With Dysphagia. The main questions it aims to answer:

Can Intermittent Nutritional Tube Supplementation help improve the nutritional status in Elderly Patients With Dysphagia.

Participants will be divided into two groups randomly. All patients are given routine rehabilitation and the intervention group is given Intermittent Oro-esophageal Tube Feeding once a day.

DETAILED DESCRIPTION:
The current situation of dysphagia in elderly individuals is characterized by difficulty or discomfort in swallowing. This condition can occur due to various factors such as muscle weakness, neurological disorders, or structural abnormalities in the throat or esophagus. Dysphagia can lead to complications such as malnutrition, dehydration, aspiration pneumonia, and reduced quality of life. It is important for healthcare professionals to assess and manage dysphagia in elderly patients to ensure proper nutrition and prevent potential health risks.

This is a prospective, randomized controlled clinical trail involved Elderly Patients With Dysphagia.The goal of this clinical trial is to compare the clinical effect of Intermittent Oro-esophageal Tube Feeding in Elderly Patients With Dysphagia. The main questions it aims to answer:

Can Intermittent Nutritional Tube Supplementation help improve the nutritional status in Elderly Patients With Dysphagia.

Participants will be divided into two groups randomly. All patients are given routine rehabilitation and the intervention group is given Intermittent Oro-esophageal Tube Feeding once a day.

ELIGIBILITY:
Inclusion Criteria:

* Age>60 years.
* Dysphagia confirmed by Videofluoroscopic Swallowing Study.
* Clear consciousness.
* Stable vital signs.

Exclusion Criteria:

* Complicated with severe liver and kidney failure, tumors, or hematological disorders.
* Simultaneously in need to undergo other therapy that might affect the outcomes of this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Nutritional status-prealbumin | Day 1 and day 15
  The relevant indicators include prealbumin (PA, mg/L) from the blood test within 24h after admission and the last day of treatment, generally, with empty-stomach ones and in the morning.

SECONDARY OUTCOMES:
Nutritional status-albumin | Day 1 and day 15
  The relevant indicators include albumin (ALB, g/L)from the blood test within 24h after admission and the last day of treatment, generally, with empty-stomach ones and in the morning.
Nutritional status-hemoglobin | Day 1 and day 15
  The relevant indicators include hemoglobin (Hb, g/L)from the blood test within 24h after admission and the last day of treatment, generally, with empty-stomach ones and in the morning.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Wi, Study Chair — Site Coordinator of United Medical Group located in Miami